CLINICAL TRIAL: NCT04173728
Title: Study of Metabolic Homeostasis in Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAS-MH-201911
Record Dates: First submitted 2019-11-07; First posted 2019-11-22 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Healthy; Metabolic Syndrome
Keywords: Metabolic health; MMTT; Resilience
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized mixed macronutrients tolerance test (Other): Subjects with different age and BMI will be included. 1) 20 subjects aged 20-29 years with normal body weight (18.5 ≤BMI<24kg/m2); 2) 40 20 subjects aged 30-70 49 years with normal body weight (18.5 ≤ BMI<24kg/m2); 3) 40 20 subjects aged 30-70 49 years with overweight or obesity (BMI<24kg/m2).); 4) 20 subjects aged 50-70 years with normal body weight (18.5 ≤ BMI<24kg/m2); 5) 20 subjects aged 30-49 years with overweight or obesity (BMI<24kg/m2); 6) 20 subjects aged 30-70 years with MetS.
  Interventions: Other: Standard mixed macronutrients tolerance test

INTERVENTIONS:
Other: Standard mixed macronutrients tolerance test — Consumption a standard mixture containing 75g glucose, 60g fat and 20 protein.

SUMMARY:
In this open-label, acute intervention study, we will recruit 120 sex-matched participants aged 20-70 years (100 normal or overweight/obese subjects and 20 Mets subjects). They will be assigned to one of the six groups according to age, BMI and with and without MetS and have a standardized mixed macronutrient tolerance test (MMTT) by orally administered a 400-ml beverage (75g glucose, 60g lipid, and 20g protein). Fasting and postprandial blood, and urine and fecal samples will be collected. The primary aim is to establish a more comprehensive system to quantify different aspects of metabolic health based on fasting and postprandial data. The study protocol has been approved by the Ethics Committee of Shanghai Institutes for Biological Sciences.

DETAILED DESCRIPTION:
The recruited 120 subjects (60 men and 60 women aged 20-70 years) will be recruited according to the followings: 1) individuals aged 20-29 years with normal weight (18.5 kg/m2 ≤ BMI < 24 kg/m2); 2) individuals aged 30-49 years with normal weight; 3) individuals aged 30-49 years with overweight/obesity (BMI ≥ 24 kg/m2); 4) individuals aged 50-70 years with normal weight; 5) individuals aged 50-70 years with overweight/obesity; and 6) individuals aged 30-70 years with MetS. A standard questionnaire will be use to collect Information like lifestyle factors, nighttime sleep duration; anthropometric measurements will be performed. Blood samples will be collected via a catheter at fasting state (t = 0 min) and 5 successive time points post-MMTT (t = 30, 60, 120, 180 and 240 min). At t = 0 ,1 and 2 h, the fingertip blood will be collected as well. Body composition will be measured by dual energy x-ray absorptiometry (DXA). All these samples will be used to the assessment of blood chemistry, metabolomics, single nucleotide polymorphism (SNP), gut microbiota etc.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects: age 20-70 BMI ≥ 18.5 kg/m2
* Mets subjects:

age 30-70 BMI ≥ 18.5 kg/m2 and at least meet three of the following criterions(NCEP-ATPIII, for Asian Americans)

1. Waist circumference ≥ 90 cm (men), ≥ 80 cm (women).
2. Total triglyceride ≥ 1.7 mmol/L.
3. HDL-c <1.03 mmol/L in men, <1.3 mmol/L in women.
4. Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg.
5. Fasting plasma glucose ≥ 5.6 mmol/L.

Exclusion Criteria:

1. clinically diagnosed diabetes or use of anti-diabetic medications;
2. clinically diagnosed cardiovascular, kidney, liver, pituitary, alimentary tract, and thyroid diseases, cancer(s), or mental illnesses;
3. pregnancy or lactation;
4. having gastrointestinal surgery within 1 year, excepting appendicitis or hernia;
5. current use of antidepressant(s);
6. alcohol consumption > 40 g/d or other substance abuse;
7. severe diarrhea (watery stools ≥ 3 times/day ≥ 3 days or longer) in previous 3 months;
8. participating any other studies within previous 3 months.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Health state map (HSM) | fasting (t = 0 min), postprandial (t = 30, 60, 120, 180, 240 min)
  A two-dimensional system comprising "Health Phenotype Score" for fasting features and "Homeostatic Resilience Score" for post-MMTT features will be built. We want to investigate whether HSM is more informative than a one-dimensional model with fasting data and the Mixed-score model combining fasting and postprandial data. Features includes BMI, blood pressure, HbA1c, body compositions, glucose, insulin, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triacylglycerol, alanine aminotransferase, aspartate aminotransferase, gamma- glutamyl transpeptidase, C-reactive protein, free triiodothyronine, free thyroxine, thyroid stimulating hormone, gastric inhibitory polypeptide, glucagon-like peptide-1, adiponectin, leptin, intercellular cell adhesion molecule-1, vascular cell adhesion molecule-1, inflammatory factors (such as interleukin, -6, -8 and 1b, and tumor Necrosis Factor-α), and targeted metabolites (such as amino acids, acylcarnitines).

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Shanghai Institute of Nutrition and Health, Chinese Acadamy of Sciences
Locations (1):
- Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China